CLINICAL TRIAL: NCT00764166
Title: Non-Metastatic High-Risk Prostate Cancer Patients With Biochemical Relapse Only After Local Treatment. A Prospective Randomized Phase III Study Comparing Hormonal Therapy +/-Docetaxel
Brief Title: A Prospective Randomized Phase III Study Comparing Hormonal Therapy +/-Docetaxel
Acronym: RisingPSA
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: ARTIC group (oncologists and urologists association) (Unknown)
Responsible Party: Aurélie Guimfack, Department Clinical Research of Developpement
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AOM 03108
Record Dates: First submitted 2008-09-30; First posted 2008-10-01 (Estimated); Last update posted 2008-10-01 (Estimated); Status verified 2008-09

CONDITIONS: Adenocarcinoma of the Prostate
Keywords: PSA (biochemical); Progression- free Survival; Clinical progress; Overall survival; Tolerance to the treatment; Quality of Live
MeSH Terms: conditions — Salivary Gland Adenoma, Pleomorphic | interventions — Docetaxel; Gonadotropin-Releasing Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Docetaxel + hormonal treatment (LH-RH agonist)
- 2 (Active Comparator)
  Interventions: Drug: Hormonal treatment (LH-RH agonist)

INTERVENTIONS:
Drug: Docetaxel + hormonal treatment (LH-RH agonist) — Docetaxel will be administered:
  * To D1 of every cycle in the dose of 70 mg/m²,
  * Perfusion IV of 60 minutes diluted in 250 ml with physiological serum or with serum glucoside from a peripheral or central vein, Every 3 weeks during 6 cycles (except when unacceptable tolerance).
  Triptorelin was given by injection for 4 times every 3 months Bicalutamide was given at the same time with LH-RH agonist for 3 weeks ; taken orally
  Arms: 1
Drug: Hormonal treatment (LH-RH agonist) — Triptorelin was given by injection for 4 times every 3 months. Bicalutamide given at the same time with LH-RH agonist for 3 weeks ; taken orally.
  Arms: 2

SUMMARY:
The primary objective was to evaluate the PSA (biochemical) progression-free survival (PFS) of high-risk metastasis-free PC patients, treated with LH-RH agonist for one year with or without docetaxel after prior radical prostatectomy (RP) or radiotherapy (RT).

The study was powered at 80% to detect a 25% improvement in biochemical PFS for a total sample size estimated at 252 patients, with a two-sided type I error rate of 5% (non-parametric methods.

DETAILED DESCRIPTION:
Docetaxel was shown to be active in metastatic hormone-refractory prostate cancer (PC) in phase III trials (1-2). It is likely to demonstrate a substantial role in the management of early-stage PC patients in the neoadjuvant and adjuvant settings, where clinical trials are underway.•53% of all men who undergo radical prostatectomy will develop prostate-specific antigen (PSA) elevations in the 10 years following surgery, with approximately 77% of these recurrences occurring within the first 2 years.A prospective, multicenter, national, randomized, two-arm, phase III study comparing hormonal treatment (LH-RH agonist alone) with or without docetaxel was designed to evaluate the interest of chemotherapy in non-metastatic prostate cancer patients at high risk of systemic recurrence after initial treatment (radical prostatectomy or radiotherapy).

1. PETRYLAK DP, et al: Docetaxel and estramustine compared with mitoxantrone and prednisone for advanced refractory prostate cancer. N Engl J Med 351:1513-1520, 2004
2. TANNOCK IF, de Wit R, Berry WR, et al: Docetaxel plus prednisone or mitoxantrone plus prednisone for advanced prostate cancer. N Engl J Med 351:1502-1512, 2004

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented adenocarcinoma of the prostate
* Previous treatment with either radical prostatectomy or radiation therapy
* Salvage radiotherapy for local relapse allowed
* Neoadjuvant or per radiotherapy Hormonal therapy allowed in case of more than 6 months free-interval before first rising PSA
* Life expectancy of more than 12 months
* Non metastatic disease documented by imaging including radionuclide bone scan
* ECOG performance status 0-1
* ANC > 1,500/mm3
* Platelet counts > 100,000/mm3
* SGOT and/or SGPT may be up to 2.5 x ULN

Patients at high risk of biological relapse defined by:

* Gleason > 8
* PSA-DT < 6 months
* Positive surgical margins
* PSA velocity > 0.75 ng/mL/year
* Pathological pelvic lymph nodes involvement (pN+)
* Time from initial treatment until inclusion < 12 months

Exclusion Criteria:

* Prior chemotherapy by taxanes and estramustine phosphate
* Documented local recurrence of prostate cancer or documented metastatic disease
* History of other malignancy within the last 5 years other than curatively treated basal cell carcinoma of the skin
* Active infection
* Significant cardiac disease, angina pectoris or myocardial infarction within twelve months
* Clinically significant neuropathy
* Medical condition requiring the use of concomitant corticosteroids
* Prohibited concomitant therapy with experimental drug.
* Participation in another clinical trial for the period < 30 days

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Actual)
Dates: Start 2003-06; Primary Completion 2009-11 (Estimated); Study Completion 2010-11 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint was the PSA (biochemical) progression-free survival (PFS) of high-risk metastasis-free PC patients, treated with LH-RH agonist for one year with or without docetaxel after prior radical prostatectomy (RP) or radiotherapy (RT). | Every month during 5 years.

SECONDARY OUTCOMES:
Secondary endpoints were metastasis-free survival, PSA response (decrease > 50 % of the PSA), overall survival, cancer specific survival, safety and quality of life (QoL). | Every month during 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Stephane Oudard, MD PhD, Principal Investigator — European Georges Pompidou Hospital
Locations (1):
- Service Oncologie Médicale, Hopital Europeen Georges Pompidou, Paris, France

REFERENCES:
- [Derived] Oudard S, Latorzeff I, Caty A, Miglianico L, Sevin E, Hardy-Bessard AC, Delva R, Rolland F, Mouret L, Priou F, Beuzeboc P, Gravis G, Linassier C, Gomez P, Voog E, Muracciole X, Abraham C, Banu E, Ferrero JM, Ravaud A, Krakowski I, Lagrange JL, Deplanque G, Zylberait D, Bozec L, Houede N, Culine S, Elaidi R. Effect of Adding Docetaxel to Androgen-Deprivation Therapy in Patients With High-Risk Prostate Cancer With Rising Prostate-Specific Antigen Levels After Primary Local Therapy: A Randomized Clinical Trial. JAMA Oncol. 2019 May 1;5(5):623-632. doi: 10.1001/jamaoncol.2018.6607. PMID 30703190